CLINICAL TRIAL: NCT07147075
Title: Provider Skill Building for Engagement and Communication in Healthcare - Hypertension Management (REACH - Hypertension)
Brief Title: Provider Skill Building for Engagement and Communication in Healthcare - Hypertension Management
Acronym: REACH - HTN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00115680; R34HL174728 (NIH)
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-08

CONDITIONS: Patient-centered Care
Keywords: Clinician Training; Patient-Centered Care; Health Equity; Hypertension Management; Pilot Trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinicians (Experimental): Doctors will complete the program over 5-6 weeks, requiring a total of 3 hours.
  Interventions: Other: REACH - Hypertension
- Patients (No Intervention): Enrolled patients will be asked to audio-record their clinical encounter with their enrolled primary care provider and complete two surveys. No intervention will be administered to the enrolled patients.
- EHR (Electronic Health Record) Cohort (No Intervention): EHR data will be collected on all patients of enrolled doctors. These patients will not consent, and no Intervention will be administered

INTERVENTIONS:
Other: REACH - Hypertension — The intervention is a skills training program for doctors that includes 3 self-paced on-line learning modules and 3 coaching sessions (one in-person and 2 virtual).
  Arms: Clinicians

SUMMARY:
Brief Summary:

The study has three main goals: The first goal is to make a skills training program that improves how doctors talk with, listen to, and work with patients. The second goal is to make sure the process of collecting data and completing the program can be done. The third goal is to make sure the skills training program is feasible and acceptable for doctors.

Study Activities:

* Doctors will first complete a questionnaire and have their patients' appointments audio-recorded.
* Then they will go through the training program.
* After finishing the program, doctors will have more patient appointments audio-recorded.
* Then the doctors will complete questionnaires again and have an interview with the study team.

ELIGIBILITY:
Inclusion Criteria:

* Doctor Cohort: Independently practicing physicians (MD, DO, PA, or NP)
* Doctor Cohort: Responsible for a panel of primary care adult patients in the Duke Primary Care clinic
* Patient Cohort: Receiving primary care from an enrolled DPC clinician at the enrolled DPC clinic
* Patient Cohort: Age at least 18 years
* Patient Cohort: Diagnosis of hypertension based on EHR ICD coding
* Patient Cohort: Able to complete a primary care encounter without an interpreter
* Patient Cohort: Able to use the study tablet for consent, data collection, and audio-recording a clinical encounter
* Patient Cohort, post-intervention: Not previously enrolled at any other timepoint
* EHR Cohort: Non-urgent patient encounters for enrolled clinicians 6 months pre intervention to 6 months post intervention completion

Exclusion Criteria:

* Doctor Cohort: Not an independently practicing physician (MD, DO, PA, or NP) at the enrolled Duke Primary Care clinic
* Patient Cohort: Previously enrolled at any other timepoint
* EHR Cohort: Urgent patient encounters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention as measured by Clinician enrollment | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
Feasibility of the intervention as measured by Patient enrollment | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
Feasibility of the intervention as measured by number of participants with completion of analyzable audio-recorded encounters | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
Feasibility of the intervention as measured by the number of participants with intervention completion | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
Feasibility of the intervention as measured by the number of participants with survey completion | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
Feasibility of the intervention as measured by the number of participants with usable electronic health record (EHR) data | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
Change in patient-centeredness as measured by Roter interaction analysis system (RIAS) | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
  Primary outcome for audio-recorded clinical encounters, the primary outcome is change in patient-centeredness, which includes behaviors like exploring the patient's perspective, showing empathy, and involving the patient in decision-making. This measure will be assessed using the Roter interaction analysis system (RIAS), a method for coding medical dialogue. The system codes each utterance (the smallest meaningful unit of speech) into one of approximately 40 categories related to task-focused or socioemotional communication. The scores derived are typically percentages or frequencies of specific communication behaviors within a given interaction (e.g., percentage of doctor talk, patient questions, or empathetic statements). A higher score is generally associated with more patient-centered communication.
Change in systolic blood pressure | Baseline - [spanning 6 months pre-intervention for all patients of the enrolled clinicians] to end point - [spanning 6 months post-intervention for all patients of the enrolled clinicians]
  A lower (mean) systolic blood pressure may suggest the intervention was effective.

SECONDARY OUTCOMES:
Change in diastolic blood pressure | Baseline - [spanning 6 months pre-intervention for all patients of the enrolled clinicians] to end point - [spanning 6 months post-intervention for all patients of the enrolled clinicians]
  A lower (mean) diastolic blood pressure may suggest the intervention was effective.
Change in hypertension control as defined by Healthcare Effectiveness Data and Information Set (HEDIS) criteria | Baseline - [spanning 6 months pre-intervention for all patients of the enrolled clinicians] to end point - [spanning 6 months post-intervention for all patients of the enrolled clinicians].
  Secondary Outcomes for EHR data is hypertension control defined by Healthcare Effectiveness Data and Information Set (HEDIS) criteria. HEDIS criteria are grouped into six domains: Effectiveness of Care, Access/Availability of Care, Experience of Care, Utilization and Risk Adjusted Utilization, Health Plan Descriptive Information, and Measures Reported Using Electronic Clinical Data Systems. HEDIS measures are used to evaluate performance on important dimensions of care and service, and are crucial for quality improvement and value-based care initiatives. A high score may suggest the intervention was effective.
Change in treatment intensification | Baseline - [spanning 6 months pre-intervention for all patients of the enrolled clinicians] to end point - [spanning 6 months post-intervention for all patients of the enrolled clinicians]
  Secondary Outcome for EHR data is treatment intensification (a measure of therapeutic inertia). These scores are calculated by comparing observed medication changes with expected changes, often based on clinical guidelines or individual patient needs. These scores range from -1 to +1. A score of 0 indicates perfect responsiveness to treatment goals, while -1 represents complete neglect, and +1 suggests excessive aggression in treatment adjustments.
Change in verbal dominance as measured by Roter interaction analysis system (RIAS) | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
  Secondary outcome for audio-recorded encounters is verbal dominance. This measure will be assessed using the Roter interaction analysis system (RIAS), a method for coding medical dialogue. The scores derived are typically percentages or frequencies of specific communication behaviors within a given interaction. The RIAS defines verbal dominance as a reflection of the patient's overall participation in the consultation, measured by their total speech time in relation to the physician's speech time. Greater change scores may suggest the intervention was effective.
Change in story questions as measured by Roter interaction analysis system (RIAS) | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
  Secondary outcome for audio-recorded encounters is story questions (lifestyle and psychosocial topics queried by the clinician). This measure will be assessed using the Roter interaction analysis system (RIAS), a method for coding medical dialogue. The scores derived are typically percentages or frequencies of specific communication behaviors within a given interaction. Greater change scores may suggest the intervention was effective.
Change in partnering behaviors as measured by Roter interaction analysis system (RIAS) | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
  Secondary outcome for audio-recorded encounters is partnering behaviors such as fostering active participation and collaboration with patients. This measure will be assessed using the Roter interaction analysis system (RIAS), a method for coding medical dialogue. The scores derived are typically percentages or frequencies of specific communication behaviors within a given interaction. Greater change scores may suggest the intervention was effective.
Change in emotional statements as measured by Roter interaction analysis system (RIAS) | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
  Secondary outcome for audio-recorded encounters is emotional statements. These measure will be assessed using the Roter interaction analysis system (RIAS), a method for coding medical dialogue. The scores derived are typically percentages or frequencies of specific communication behaviors within a given interaction. Greater change scores may suggest the intervention was effective.
Change in encounter duration as measured by Roter interaction analysis system (RIAS) | Baseline (pre-intervention), within 6 weeks post-intervention, and 12-16 weeks post-intervention
  Secondary outcome for audio-recorded encounters is encounter duration. This measure will be assessed by the length of the recorded dialogue of the Roter interaction analysis system (RIAS), a method for coding medical dialogue. Longer recorded encounters may suggest the interventon was effective.

CONTACTS AND LOCATIONS:
Overall Officials: Investigator, PhD, Principal Investigator — Duke University; Investigator, MD, Principal Investigator — Duke University
Locations (1):
- Duke Primary Care South Durham, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual Particpant Data (IPD) will not be shared

DOCUMENTS (3):
  • Informed Consent Form: Clinician (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/75/NCT07147075/ICF_000.pdf
  • Informed Consent Form: Patient (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT07147075/ICF_001.pdf
  • Informed Consent Form: 3rd party (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT07147075/ICF_002.pdf